CLINICAL TRIAL: NCT01047150
Title: The Comparison of the Necessity of Repeat Myocardial Perfusion SPECT Studies Between Tc-99m Tetrofosmin and Tc-99m Sestamibi
Brief Title: The Comparison of the Necessity of Repeat Myocardial Perfusion SPECT Studies Between Tc-99m Tetro and Tc-99m Mibi
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cardiac Imaging of Augusta (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Gordon Leslie Walters, MD, Cardiac Imaging of Augusta
Other Study IDs: DB1
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-12

CONDITIONS: Myocardial Ischemia
Keywords: Myocardial Perfusion Imaging; Repeat studies; Tetrofosmin; Sestamibi
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Tetrofosmin Rest patients: Patients that had a Rest myocardial perfusion study using Tc99m tetrofosmin
- Sestamibi stress patients: Patients that had a stress myocardial perfusion imaging study using Tc99m Sestamibi
- Tetrofosmin stress patients: Patients that had a stress myocardial perfusion imaging study using Tc99m Tetrofosmin
- Sestamibi rest patients: Patients that had a rest myocardial perfusion imaging study using Tc99m Sestamibi

SUMMARY:
Research Questions:

1. Is there a significant difference between the causal repeat rate of myocardial perfusion studies for Tc99m tetrofosmin and Tc99m sestamibi?
2. Is there a significant difference in the causal repeat rate of myocardial perfusion studies for Tc99m tetrofosmin and Tc99m sestamibi if an independent technologist reviewer blinded to the radiopharmaceutical makes the decision to repeat the study?
3. Is there a significant difference in the quantitative diagnostic measures reported between the original and the acceptable repeated studies?

DETAILED DESCRIPTION:
There are two commonly used Tc-99m based radiopharmaceuticals useful in the diagnosis and localization of regions of reversible myocardial ischemia in the presence or absence of infarction under exercise and rest conditions. One is Tc-99m tetrofosmin (Tc-99m-1,2-bis[bis(2-ethoxyethyl) phosphino] ethane), the other is Tc-99m sestamibi (Tc-99m- methoxyisobutylisonitrile). When performing a myocardial perfusion SPECT (MPS) study, extracardiac subdiaphragmatic activity adjacent to the myocardium can cause artifacts in the inferior wall and can be detrimental to the accuracy of the study1,2. Following acquisition, MPS studies are routinely checked for potential imaging artifacts. When a separation between the extracardiac activity cannot clearly be distinguished from the myocardium, the study should be repeated. Repeating the SPECT study can affect the efficiency of a lab as well as having a negative influence on patient comfort and overall satisfaction. The goal of this study is to determine if there is a significant difference in the number of studies that should be repeated between the two commonly used radiopharmaceuticals.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving sestamibi MPI study or tetrofosmin MPI study

Exclusion Criteria:

* Thallium or dual isotope MPI study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for MPI
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Number of studies repeated. | four weeks

SECONDARY OUTCOMES:
Number of studies that should have been repeated | two weeks after data collection

CONTACTS AND LOCATIONS:
Overall Officials: Danny A Basso, CNMT, Study Director — Cardiac Imaging of Augusta
Locations (1):
- Cardiac Imaging of Augusta, Augusta, Georgia, United States